CLINICAL TRIAL: NCT01068171
Title: Developing a Diabetic Foot Ulcer Protocol in a Multi-ethnic, Underserved Population
Brief Title: Developing a Diabetic Foot Ulcer Protocol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients who met enrollment criteria
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Harris County Hospital District (Other Government); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-GEN-09-0418
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: diabetes; foot ulcers; off-loading; collagen; Wagner 1
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — Silver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- shoe, plain dressing (Active Comparator): post-op shoe with plain occlusive dressing
  Interventions: Other: type of footwear
- shoe, collagen (Active Comparator): post-op shoe with collagen dressing
  Interventions: Other: collagen dressing with and without silver
- boot, plain dressing (Active Comparator): air boot with occlusive dressing
  Interventions: Other: type of footwear
- boot, collagen (Active Comparator): air boot with collagen dressing
  Interventions: Other: collagen dressing with and without silver
- monitored air boot, plain dressing (Active Comparator): air boot with retention strap to monitor whether boot is removed with occlusive dressing
  Interventions: Other: type of footwear
- monitored boot with collagen (Active Comparator): air boot with retention strap to monitor whether boot is removed with collagen dressing
  Interventions: Other: collagen dressing with and without silver

INTERVENTIONS:
Other: type of footwear — comparison of results between post-op shoe, air boot which the patient can remove ad lib and air boot whose removal can be monitored
  Other Names: DJO XP Diabetic Walker; Camcon Medical postoperative shoe; Smith and Nephew Allevyn Foam dressing
  Arms: boot, plain dressing; monitored air boot, plain dressing; shoe, plain dressing
Other: collagen dressing with and without silver — silver-impregnated collagen dressing will be used for 2 weeks, then plain collagen dressing will be used for the remainder of the 6 months
  Other Names: Smith & Nephew Biostep dressing with Allevyn Foam cover; Smith & Nephew Biostep Ag gressing with Allevyn Foam cover
  Arms: boot, collagen; monitored boot with collagen; shoe, collagen

SUMMARY:
The purpose of this study is to determine which treatment, over 6 months, will promote healing of diabetic foot ulcers that are not infected in the most efficient, cost-effective way.

DETAILED DESCRIPTION:
This pilot study will be conducted in Harris County Hospital District (HCHD) Community Health Centers and Wound Care Clinics.

The study will use random assignment of patients who meet inclusion criteria to: postoperative shoe with or without collagen; removable Air-boot with or without collagen; or monitored Air-boot with or without collagen. All treatment is standard of care.

Enrollment will occur at a clinic appointment. During the consent appointment, follow-up will be scheduled. Patients whose wound meets study criteria will be approached by a Podiatrist or therapist during a wound care visit. An A1c will be obtained, if not done within the past 3 months. A convenience sample will be drawn from people with diabetes, aged 18 or more, who meet inclusion criteria.

Frequency of visits will be:

* patients with monitored Air-boot: weekly
* all others: every 2 weeks At each visit there will be a dressing change, wound assessment and review of how many times shoe/boot was removed or not used during the preceding 1 or 2 weeks.

Should healing not occur within 6 months or the wound progress, the patient will be referred for evaluation of possible vascular involvement.

ELIGIBILITY:
Inclusion Criteria:

* Adult - over 18 years of age
* Diabetes with an A1c of less than or equal to 9% - if no A1c result is available within the past 3 months, one will be drawn to qualify the patient for the study
* No evidence of circulatory compromise

  * Posterior tibial or pedal pulse present on palpation
  * No pallor on elevation
  * No dependent rubor
* Loss of sensation on forefoot using monofilament
* Wound or callus on only 1 foot
* Wound Classification - Wagner Grade 1, non-infected

  * Ulcer present for 1 - 3 months
  * Ulcer of forefoot only
  * No previous ulcer of that foot or amputation of either extremity
  * Wound size < 1" diameter
  * Wound bed pink

Exclusion Criteria:

* Diagnoses with unpredictable trajectory or healing ability, i.e.

  * Psychiatric disorders
  * Cancer
  * ESRD not eligible for dialysis
  * HIV
* Previous lower extremity amputation
* Charcot foot
* Evidence of circulatory compromise

  * Absence of pulses
  * Decreased capillary refill (> 3 seconds)
  * Trophic skin changes - shiny, hairless toes
  * Ankle Brachial Index < 0.8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
decrease in size of wound | 6 months

SECONDARY OUTCOMES:
non-healing wound | 6 months or less

CONTACTS AND LOCATIONS:
Overall Officials: Gary Lepow, DPM, Principal Investigator — University of Texas Health Science at Houston, Baylor College of Medicine; Talar L Glover, MS, RN, CNS, Principal Investigator — Harris County Hospital District
Locations (1):
- Harris County Hospital District Community Health, Houston, Texas, United States